CLINICAL TRIAL: NCT02591134
Title: SWITCH: EffectS of Non-nutritive sWeetened Beverages on appetITe During aCtive weigHt Loss
Brief Title: EffectS of Non-nutritive sWeetened Beverages on appetITe During aCtive weigHt Loss
Acronym: SWITCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Jason Halford (Other)
Collaborators: American Beverage Association (Other)
Responsible Party: Sponsor-Investigator, Professor Jason Halford, Professor, University of Liverpool
Organization: University of Liverpool (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ULKLABA01
Record Dates: First submitted 2015-10-23; First posted 2015-10-29 (Estimated); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Weight
Keywords: weight loss; NNS; beverages; diet; appetite; satiety; weight control
MeSH Terms: conditions — Body Weight; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non Nutritive Sweetened Beverages (Experimental): Non-nutritive sweeteners (NNS) beverages will be provided to participants using a home delivery system and they are expected to consume at least two portions (330ml) per day.
  Interventions: Other: Non Nutritive Sweetened Beverages
- Control Water Beverages (Placebo Comparator): Water beverages will be used as a comparator to NNS beverages during the trial. These beverages will encompass a range of water-based drinks that contain no NNS. Including water as a comparator is vital to understand whether NNS beverages are equally as effective as water during phases of weight loss and weight maintenance.
  Interventions: Other: Control

INTERVENTIONS:
Other: Non Nutritive Sweetened Beverages — Non-nutritive sweeteners (NNS) beverages encompass a range of carbonated and still drinks with added artificial sweeteners. Participants will be provided with a list of permitted beverages and are expected to consume at least two portions (330ml) per day.
  Arms: Non Nutritive Sweetened Beverages
Other: Control — Water beverages provided in 330ml portions to be consumed twice per day over the duration of the trial
  Arms: Control Water Beverages

SUMMARY:
The effects of non-nutritive sweetened (NNS) beverages on weight management and psychological indices of appetitive behaviour have not been assessed in both weight loss and maintained weight loss phases over the long term to determine whether NNS beverages may assist in efforts to lose weight and maintain weight loss and how this affects appetite expression (satiety, food choice, craving, ease of dieting etc.). Thus the present research will determine the impact of NNS beverages as compared to water on weight loss and weight loss maintenance, satiation, satiety, cravings for sweet, exercise efforts and mood state across both a period of weight-loss as well as a weight-maintenance phase. To determine if the effects of NNS on appetite are beneficial or detrimental to successful weight management, the study will also systematically compare the effects of NNS beverages, water and caloric beverages (CBs) on appetite (hunger, satiety, liking and wanting) and energy intake (including food choice and caloric compensation) across the whole day during active weight management in a subset of participants.

DETAILED DESCRIPTION:
The study will use a parallel randomized design with two arms; participants will either be randomized to a non-nutritive sweetener (NNS) beverage condition (active) or a water condition (control). A total of 432 overweight and obese participants (Body Mass Index; BMI range: 27-35 kg/m2) will be enrolled in the study. A 3-month weight loss diet phase will initially be completed, with participants receiving nutritional advice at weekly group sessions whilst additionally incorporating the active or control products into their diet (weeks 0-12). This programme is based on a model successfully used in an American sample (Peters et al., 2014) which will be adapted for a UK sample. This will be followed by a 9-month weight maintenance phase (weeks 13-49) in which participants will be advised to follow a general healthy diet in accordance with dietary guidelines (continuing to incorporate the active or control beverages) but will only attend monthly group sessions. This will be followed by a voluntary one year post assisted weight maintenance period in which participants will continue to consume the active or control beverages every day and will be asked to complete questionnaire measures, cognitive tasks, biomarkers of health (blood samples, if willing) and body composition data (weight, sagittal diameter and hip and waist circumference measures; DXA (for Subset 2)) at the end of this period. A subset of participants (Subset 1) will additionally undergo appetite probe days (n = 116), attending the Study Centre at 15 points throughout the trial (3 sessions at baseline, 3 sessions at the start of the weight loss programme, 3 sessions at the end of the weight loss programme, 3 sessions at the end of assisted weight maintenance and 3 sessions at the end of the one year post assisted weight maintenance period). A separate subset (Subset 2) will complete biological assessment measures (n =50) involving body composition (DXA) scans at 4 points throughout the trial (at baseline, end of weight loss, end of assisted weight maintenance, and at a year post assisted weight maintenance visit) and all participants will be asked to provide blood samples at these four points but will not be excluded from the trial should they not wish to.

Both groups will be asked to ensure that they consume at least two servings (330 ml) of their elected beverages dependent on condition (NNS vs. water). All beverages will be picked by participants (from a permitted range) and then delivered to them in bi-weekly batches using an online delivery-style system. Primary study visits for body weight, waist circumference, hip circumference, sagittal diameter, and blood pressure assessments will be carried out at various stages throughout the trial. Initial assessments will be at baseline (week -2), monthly over the weight loss period (weeks 4, 8 and 12), monthly over the assisted weight maintenance period (weeks 16, 20, 24, 28, 32, 36, 40, 44 and 48) and at a 1 year post assisted weight maintenance visit with Subset 2 additionally providing body composition (DXA) scans at baseline, at the end of the weight loss period, at the end of the assisted weight maintenance period and at a 1 year post assisted weight maintenance visit. During the weight loss phase, participants will meet in groups (10-12 participants) with a dietician-trained researcher every week (12 visits) followed by monthly meetings during the assisted weight maintenance phase (9 visits). Participants will additionally be asked to complete a series of questionnaires throughout the intervention period and complete a series of diet diaries (3-day diet diaries and food frequency questionnaires; FFQs) to assess compliance throughout the trial. Furthermore, empty product packaging (labels or bottles) will be collected as an additional compliance measure. The probe days to be completed by Subset 1 will involve participants attending the Study Centre at various times over an 8-hour day period for 3 meals (breakfast, lunch and dinner) and 1 drink (NNS, sugar sweetened beverage (SSB) or water) for a total of 15 sessions. Adverse events and concomitant medicine will be registered continuously throughout the study in relevant forms. For each participant, the total study duration is 100 weeks (not including recruitment and screening but including the voluntary post assisted weight maintenance phase) and includes a total of 39 visits (with additional visits for Subsets 1 and 2).

12-week weight loss programme. The 12-week Weight Loss Programme (WLP) will be based on the current successful UK-based dietician-designed nutritional knowledge and group work programme used within the Kissileff Laboratory, the content of which will be enhanced by a social cognition based programme currently used in Colorado. This employs a group based approach (10-12 participants) with frequent meetings (one per week) for a one hour session with a dietician trained researcher who will supervise the sessions and who will provide materials and 'home work' for the participants to complete before their next session. This programme will be tailored for the UK and specific behavioural components such as advice on self-monitoring, stimulus control, stress management, slow eating rate and related behaviours will be covered. An exercise component will also be included in which exercise activities are noted in a log and an additional online daily drinking log will also be included. The exercise log will be completed weekly and brought to each session as a means of monitoring. Weight will be measured at the start and end of this phase and weekly during the WLP as part of group sessions (at the end of the group session) and will be conducted privately with each participant in a separate room. Participants will also be asked to complete food frequency questionnaires (FFQs) once per month and online 3-day diet diaries before beginning the WLP and at the end of the WLP and will be given instructions on how to do so. In week 12 a further visit (independent from group sessions) will be scheduled individually with each participant to complete additional questionnaire and cognitive measures (Visit 13).

36-week assisted weight maintenance phase. Participants will be asked to attend one hour monthly group sessions with a dietician-trained researcher (10-12 participants per group) during the 36-week assisted weight maintenance phase running from week 13-48. These meetings will provide an opportunity for participants to discuss any concerns and to provide further reminders of nutritional advice. Body weight will be measured at the end of each group session and will be conducted privately with each participant in a separate room. Participants will also be asked to complete a series of questionnaires measuring appetite control and ease of dieting and measures of dietary compliance alongside providing the online daily beverage log and weekly paper exercise log. Participants will also be asked to complete FFQs monthly during this period. At the end of this phase further visits (independent from group sessions) will be scheduled to complete the final measures of appetite and food choice and to provide their final online 3-day diet diary.

Fasting blood samples will be analysed for glucose, insulin, lipids, triglycerides, high density lipoprotein (HDL), low density lipoprotein (LDL), total cholesterol profiles and Hba1.

One year post assisted weight maintenance and visit After the final study visit post-maintenance (week 48), participants will continue to be provided either NNS or water beverages for a 12-month duration. They will be asked to return their empty beverage packaging monthly during this phase (weeks 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96) and will complete retrospective appetite questionnaires alongside additional questionnaires upon returning their packaging. They will also complete daily online beverage logs online over the duration of the 12-month period and will complete a final online 3-day food diary which they present at Visit 39 (week 100). Participants in Subset 1 will additionally undergo a final set of probe days in weeks 98-99 (Visits 38a, 38b, and 38c). Subset 2 will also provide their final DXA scan at the one year post assisted weight maintenance period visit (Visit 39). At this final visit participants will be asked to provide a fasting blood sample as well as complete a range of computer tasks, questionnaires and food diaries. Their body weight will be measured and their waist, hip and sagittal diameter will be taken in a separate room along with their blood pressure

Subsets Subset 1 - Appetite Probe Days A voluntary subset of randomly selected participants (n=116) will be invited to participate in the appetite probe day sessions to assess changes in appetite response to caloric and non-caloric beverages (water, NNS and caloric beverages; CB). These probe days will be measured at baseline (Visits 2a, 2b & 2c; weeks -2 to 0), at the start of the weight loss programme (Visits 3a, 3b and 3c; weeks 1 to 2), at the end of the weight loss period (Visits 13a, 13b and 13c; weeks 11 to 12) at the end of the assisted weight maintenance period (Visits 24a, 24b, 24c; weeks 47 to 48) and at the end of the 1 year post assisted weight maintenance period (Visits 38a, 38b, & 38c). These sessions will be scheduled a minimum of 3 days after one another (minimum completion of 2 weeks) and must all be completed within a maximum of 3 weeks. At each point one probe day will examine the response to a caloric beverage (ie a sugar sweetened beverage; SSB) and then the second and third the response to NNS and water (the order of all three drinks will be counterbalanced across participants and probe days). These will be provided after breakfast and 1 hour before lunch (approximately 12pm). Compensation will then be tracked at an ad libitum test lunch and an evening meal. Participants will be blinded to the study condition (no information will be provided about the drinks during the probe days) however the sensory characteristics of the beverages may be evident. Cognitive and sensory cues cannot be matched but are important determinants of real world appetite responses.

The gold standard 8-hour design will be used. The appetite probe day will be conducted at the Kissileff Laboratory study centre and will involve participants attending the centre for a fixed breakfast (breakfast is calibrated based on weight bands which will be determined at the Screening session; prior to the end of WLP and prior to the end of the assisted weight maintenance phase to ensure accurate weight banding), the study beverage, ad libitum lunch and ad libitum dinner as well as a take-home snack pack for the remainder of the evening. Participants will complete appetite VAS pre- and post- each meal as well as completing these ratings at hourly intervals throughout the test day. They will be free to leave the Study Centre after consuming their meals and will be provided with water as well as a specified time to return for their next meal.

Subset 2 - DXA Scans In addition to trial participation, Subset 2 (n = 50) be asked to provide fasting full body DXA scan at dedicated visits 1d, 14a, 25a, and 39 (weeks 0, 12, 48 and the one year post assisted weight maintenance visit respectively). The DXA scan will be used to assess changes in body composition during the trial.

Participants will be reminded during the Screening session that they do not have to take part in the additional testing (Subsets 1 or 2) or provide blood samples to be eligible for enrolment in the trial.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 27.0 and ≤ 35.0 kg/m2
* Healthy
* Age between 18 and 65 years (inclusive)
* Regular consumer of cold NNS or water beverages (>3 per week but < 2 litres per day)
* Acceptance of randomization to either a water or NNS beverage condition
* Willing to abstain from consuming NNS beverages (if randomized to the water condition) and SSBs for the duration of the trial.
* Provided voluntary written informed consent
* Not planning on moving outside of the local area in the next 24 months
* Two individuals from the same household complying with the inclusion and exclusion criteria will be permitted to participate in the trial however, in such instances, the individuals will be randomized to the same group

Exclusion Criteria:

* Not willing to discontinue drinking NNS beverages for the duration of the trial should they be assigned to the water group and vice versa;
* Not willing to consume NNS beverages or water for the duration of the trial;
* Expressing a significant dislike of NNS beverages (at least moderately likeable on a 5 point likert scale);
* Excess consumer of chilled beverages or NNS beverages (more than 2 litres a day);
* A BMI below 27 or above 35 kg/m2;
* Below the age of 18 or above 65 years;
* A first year University Student (to avoid the 'freshman 15' phenomenon of weight gain within the first year of attending University);
* Significant health problems (including a history of cardiovascular diseases);
* Gastro-intestinal problems or diabetes;
* Taking any medication or supplements known to affect appetite or weight within the past month and/or during the study;
* Stated major psychiatric disorder (made clear by medicines specified);
* Current depression (made clear by medicines specified);
* Currently being treated for a psychological condition;
* Being pregnant, planning to become pregnant, breastfeeding or less than 6 months post-partum;
* Planning on moving away from the local area within the next two years;
* History of anaphylaxis to food; known food allergies or food intolerance;
* Dislike of > 25% of the study foods offered on the appetite probe day (Subset 1 only);
* Non breakfast eaters (subset 1 only);
* Smoking or having ceased smoking in the last six months;
* Currently dieting, having ceased a diet in less than 4 weeks, or having lost significant amounts of weight in the previous year;
* Engaging in regular intense exercise;
* Having significantly changed their physical activity patterns in the past 4 weeks or intending to change them during the study (other than to adhered to advice given in the behavioural intervention);
* Inability to adhere to the programme such as inability to increase activity level;
* Receiving systemic or local treatment likely to interfere with evaluation of the study parameters;
* Working in appetite or feeding-related disciplines;
* Being on specific food avoidance diets;
* Having had bariatric surgery;
* Having abnormal eating behaviour (restrained eaters measured by the Dutch Eating Behaviour Questionnaire - Restraint Scale [DEBQ-R] with a cut-off point of more than 4 (van Strien et al,1986); and binge eaters measured by the Binge Eating Scale with a cut-off point of 27 or over (Gormally et al, 1982))

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2016-07; Primary Completion 2024-02 (Actual); Study Completion 2024-02 (Actual)

PRIMARY OUTCOMES:
Initial change in weight | 52 weeks
  weighing participants (kilograms)

SECONDARY OUTCOMES:
Changes in appetite/programme experience (all VAS) | 52 weeks
  The experience of the weight loss programme and weight maintenance phases via associated questionnaires as well as assessments of appetite throughout the trial to detect changes in satiety (via associated questionnaires) - all one unit of measurement
Circulating biomarkers of health | 52 weeks
  Blood samples from all willing
Effects of beverages on food choice | 52 weeks
  Subset 1 will complete study days in which they are provided with caloric beverages, water or NNS beverages. Subsequent food choices with ad-libitum meals will then be assessed at various time points over the trial (calories consumed)
Body composition change | 52 weeks
  Anthropometric measures (DXA in Subset 2)
Waist, hip and sagittal changes | 52 weeks
  Measurements in whole sample (all in centimetres)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Halford, Professor, Principal Investigator — University of Liverpool
Locations (1):
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Ethically we cannot share individual participant data that may identify the individual. As stated in NHS ethics we do not plan on sharing this data with external parties to the PI, CI or University of Liverpool staff employed on the project

REFERENCES:
- [Background] van Strien T, Oosterveld P. The children's DEBQ for assessment of restrained, emotional, and external eating in 7- to 12-year-old children. Int J Eat Disord. 2008 Jan;41(1):72-81. doi: 10.1002/eat.20424. PMID 17634965
- [Background] Gormally J, Black S, Daston S, Rardin D. The assessment of binge eating severity among obese persons. Addict Behav. 1982;7(1):47-55. doi: 10.1016/0306-4603(82)90024-7. PMID 7080884
- [Background] Peters JC, Wyatt HR, Foster GD, Pan Z, Wojtanowski AC, Vander Veur SS, Herring SJ, Brill C, Hill JO. The effects of water and non-nutritive sweetened beverages on weight loss during a 12-week weight loss treatment program. Obesity (Silver Spring). 2014 Jun;22(6):1415-21. doi: 10.1002/oby.20737. PMID 24862170
- [Derived] Harrold JA, Hill S, Radu C, Thomas P, Thorp P, Hardman CA, Christiansen P, Halford JCG. Non-nutritive sweetened beverages versus water after a 52-week weight management programme: a randomised controlled trial. Int J Obes (Lond). 2024 Jan;48(1):83-93. doi: 10.1038/s41366-023-01393-3. Epub 2023 Oct 5. PMID 37794246
- [Derived] Masic U, Harrold JA, Christiansen P, Cuthbertson DJ, Hardman CA, Robinson E, Halford JC. EffectS of non-nutritive sWeetened beverages on appetITe during aCtive weigHt loss (SWITCH): Protocol for a randomized, controlled trial assessing the effects of non-nutritive sweetened beverages compared to water during a 12-week weight loss period and a follow up weight maintenance period. Contemp Clin Trials. 2017 Feb;53:80-88. doi: 10.1016/j.cct.2016.12.012. Epub 2016 Dec 12. PMID 27979755